CLINICAL TRIAL: NCT03406481
Title: The Impact of Preoperative Fasting Period on Cardiac Index Variability After Anesthesia Induction in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2017.669
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Fasting Period; Intravascular Volume

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The minimum period of fasting recommended by the 'American Society of Anesthesiologists' for the preoperative period is 6 hours for solid foods and 2 hours for clear liquids. Knowing the effect of preoperative fasting time on intravascular volume status may lead us to determine the amount of fluid to be administered intraoperatively. Cardiac preload static indicators are often insufficient to predict the need for fluid and are often measured by invasive methods. Knowing the adequacy of the preload is important in anesthesia practice; there is no hemodynamic benefit of fluid replacement in non-responsive patients. In this study, the investigators aimed to determine the effect of preoperative fasting period on cardiac index change after anesthesia induction in pediatric patients aged 5-12 years. The primary implication of this study is to determine the fasting period of fluid evacuation by assessing patients' intravascular volume status.

ELIGIBILITY:
Inclusion Criteria: pediatric patients, aged between 5 to 12, undergoing surgery -

Exclusion Criteria: any comorbidity

-

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: pediatric patients undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
the relationship between fasting period duration and fluid responsiveness | March 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No